CLINICAL TRIAL: NCT06132945
Title: Phase 1b Study of the Safety of Concurrent Cabozantinib and Nivolumab With Radiation Therapy for Brain Metastases in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Study of Cabozantinib and Nivolumab With Radiation Therapy for People With Renal Cell Carcinoma That Has Spread to the Brain
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-138
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Brain Metastases
Keywords: Cabozantinib; Nivolumab; Stereotactic Radiosurgery (SRS); 23-138
MeSH Terms: conditions — Carcinoma, Renal Cell; Brain Neoplasms | interventions — cabozantinib; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a single-institution, single cohort, phase 1b trial of cabozantinib in combination with nivolumab in patients with metastatic RCC who are planning to undergo radiation therapy for brain metastases.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib and Nivolumab With Radiation Therapy (Experimental): Patients being newly initiated on cabo/nivo will be started on with cabozantinib 40 mg PO daily and nivolumab 480 mg IV day Q4 weeks
  o Dose de-escalation of cabozantinib for toxicity will be allowed per prespecified toxicity dose levels
  Radiation will be stereotactic radiosurgery, delivered over 1-5 fractions with a total dose of 18-30Gy depending on fractionation schedule per the discretion of the treating radiation oncologist. Standard institutional regimens such as 18-24 Gy in a single fraction, 24-27 Gy in three fractions, and 25-30 Gy in five fractions are permissible.
  Interventions: Drug: Cabozantinib; Device: Nivolumab; Radiation: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib (40 mg PO daily)
Device: Nivolumab — Nivolumab (480 mg IV Day 1)
Radiation: Stereotactic Radiosurgery (SRS) — Radiation will be stereotactic radiosurgery, delivered over 1-5 fractions with a total dose of 18-30Gy depending on fractionation schedule per the discretion of the treating radiation oncologist.

SUMMARY:
The purpose of this study is to find out whether the combination of cabozantinib, nivolumab, and radiation therapy is a safe and effective treatment that causes few or mild side effects in people with renal cell cancer that has spread to the brain. The researches will also look at how the study treatment affects the quality of life of participants. They will measure the quality of life by having participants complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable advanced or metastatic clear cell or non-clear cell RCC; all histologies acceptable except for chromophobe RCC
2. Brain metastases present, meeting the following criteria:

   1. At least 1 brain metastasis measuring ≥0.5cm in any dimension (intracranial RANO-BM measurable disease required)
   2. SRS is indicated per treating radiation oncologist
   3. Surgical intervention for brain metastases is not planned
3. Able to undergo MRI Brain assessments for radiation planning.
4. Availability of archival tissue that enables the definitive diagnosis of RCC, accompanied by an associated pathology report. If archival tissue cannot be obtained, PI to provide documented confirmation patient can still enroll onto the study. Specimens can be collected by surgical resection or biopsy of the primary tumor or biopsy or resection of a metastatic lesion.
5. Age ≥18 years
6. KPS ≥ 80
7. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 28 days prior to the first study treatment:

   1. ANC ≥ 1500 cells/μL (without granulocyte colony stimulating factor support within 4 weeks prior to Cycle 1, Day 1)
   2. WBC counts ≥ 2500/μL
   3. Absolute lymphocyte count ≥ 500/μL
   4. Platelet count ≥100,000/μL (without transfusion within 4 weeks prior to Cycle 1, Day 1)
   5. Hemoglobin ≥9.0 g/dL o Patients may be transfused or receive erythropoietic treatment to meet this criterion.
8. AST, ALT, and alkaline phosphatase ≤ 2.5 x ULN, with the following exceptions:

   1. Patients with documented liver metastases: AST and/or ALT ≤ 5 x ULN
   2. Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
9. Serum bilirubin ≤ 1.5 x ULN
10. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be- enrolled.
11. INR and aPTT ≤ 1.5 x ULN

    a. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
12. Creatinine ≤ 1.5 x ULN or Calculated Creatinine clearance ≥ 30mL/min by institutional standard measurement
13. For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception, including at least one method with a failure rate of ≥ 1% per year
14. If any Grade ≥1 toxicities occurred in relation to prior treatment, patients must have recovered to baseline or ≤ Grade 1 unless adverse events are clinically insignificant or stable on supportive medication if needed.

Exclusion Criteria:

1. Prior treatment with cabozantinib for RCC
2. Receipt of any small molecule kinase inhibitor (including investigational) or VEGFtargeted therapy within 2 weeks before the first dose of study treatment

   o 2-week washout period was selected in order to facilitate rapid enrollment and treatment of patients given the target population with active brain metastases.
3. Patients requiring whole brain radiotherapy (WBRT).
4. Any prior brain radiotherapy within 28 days prior to enrollment
5. Incomplete healing from prior radiotherapy as determined by the treating radiation oncologist or treating investigator
6. Diagnosis of autoimmune condition that may worsen during immune checkpoint blockade, with the following exceptions:

   o Diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
7. Any active or suspected autoimmune disease requiring systemic steroids > 10 mg daily prednisone (or equivalent) or other immunosuppression, except for:

   * those not expected to reoccur
   * Chronic physiologic replacement of ≤10mg prednisone (or equivalent) for treatment of adrenal insufficiency
   * Steroids required for pre-medication reactions
   * Local steroid use is permitted (e.g. intranasal, topical, inhaled, or local steroid injection, i.e. intra-articular)
8. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
9. Uncontrolled hypercalcemia (≥ 1.5 mmol/L ionized calcium or Ca ≥ 12 mg/dL or corrected serum calcium ≥ ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
10. Participation in an experimental drug study within 28 days of study enrollment
11. Pregnant and lactating women
12. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
13. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina, or EF < 50%

    o Patients with known coronary artery disease, congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
14. Uncontrolled hypertension (>140 mm Hg systolic or >90 mm Hg diastolic) despite optimal antihypertensive treatment
15. QTcF > 500 msec within 28 days before the first dose of study treatment
16. Major surgical procedure within 14 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study

    o Patients must have completed wound healing from major or minor surgery before first dose of study treatment
17. History of stroke or transient ischemic attack within 6 months prior to Cycle 1, Day 1
18. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1
19. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)

    o Clinically significant hematuria, hematemesis, or hemoptysis of >0.5 tsp (2.5ml) of red blood or other history of significant bleeding within 12 weeks before first dose of study treatment.
20. Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
21. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
22. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
23. Concomitant anticoagulation with coumarin agents, direct thrombin inhibitors, factor Xa inhibitor betrixaban, or platelet inhibitors. Other anticoagulants are allowed.
24. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

    o Complete healing of intra-abdominal abscess must be confirmed before the first dose of study treatment
25. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
26. Lesions invading or encasing major blood vessels
27. Uncompensated or symptomatic hypothyroidism
28. History of solid organ or allogeneic stem cell transplant
29. Clinically significant active infection including HIV, Hepatitis B, Hepatitis C, acute COVID-19 infection, or other

    * For patients with HIV infection, clinically significant/exclusionary features include: detectable viral load, CD4+ T cell count <300 cells/microL, or history of opportunistic infection
    * For patients with HBV infection, clinically significant/exclusionary features include: HBV surface antigen positivity, detectable HBV DNA by polymerase chain reaction (PCR). Patients with prior HBV infection (HBV core Ab positive, HBV DNA undetectable by PCR, HBV surface antigen negative) are eligible for the study if they are already stable on entecavir or tenofovir
30. Inability to swallow tablets
31. Previously identified allergy or hypersensitivity to components of the treatment
32. Malignancy that requires anti-cancer directed therapy within the last 3 years. Exceptions include those cancers that are considered cured by local therapy (e.g. Basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of breast, bladder, or cervix) or other cancers that have low malignant potential and do not require systemic therapy (e.g. Gleason grade <6 prostate adenocarcinoma)
33. Patients in whom nivolumab treatment is not otherwise feasible (for example, for financial reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
percent of enrolled patients who are able to tolerate treatment | 56-day
  56-day safety monitoring period without unacceptable CNS toxicity. Unacceptable CNS toxicity is defined as any grade ≥3 treatment-emergent neurological disorder, per NCI CTCAE version 5.0 criteria

SECONDARY OUTCOMES:
rate of CNS adverse events | 1 year
  CNS adverse events will be reported as a proportion of patients who experience a CNS adverse event of any grade based on CTCAE 5.0
objective response rate (ORR) | 1 year
  as measured by RANO-BM criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Kotecha, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm